CLINICAL TRIAL: NCT00928226
Title: A Phase I/II Study of Fractionated Stereotactic Radiosurgery to Treat Large Brain Metastases
Brief Title: Study of Fractionated Stereotactic Radiosurgery to Treat Large Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Soltys, Assistant Professor of Radiation Oncology, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15107; SU-04272009-2418 (Other: Stanford University); BRN0010 (Other: OnCore)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Brain Cancer; Neoplasm Metastasis; Cancer of Brain and Nervous System; Metastatic Malignant Neoplasm to Brain
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Arm 1 - 24 Grey SRS (Experimental): 24 Grey administered as 8 Gy x 3 fractions
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery (SRS); Procedure: Surgical resection
- Arm 2 - 27 Grey SRS (Experimental): 27 Grey administered as 9 Gy x 3 fractions
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery (SRS); Procedure: Surgical resection
- Arm 3 - 30 Grey SRS (Experimental): 30 Grey administered as 10 Gy x 3 fractions
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery (SRS); Procedure: Surgical resection
- Arm 4 - 33 Grey SRS (Experimental): 33 Grey administered as 11 Gy x 3 fractions
  Interventions: Radiation: Fractionated Stereotactic Radiosurgery (SRS); Procedure: Surgical resection

INTERVENTIONS:
Radiation: Fractionated Stereotactic Radiosurgery (SRS) — Standard of care
  Other Names: Cyberknife surgery
Procedure: Surgical resection — Standard of care

SUMMARY:
The maximum tolerated dose of 3-session (ie, treatment) stereotactic radiosurgery (SRS) to treat brain metastases greater than 4.2 cm³ in size will be determined.

This study investigates if increasing radiation dose improves outcome for patients without greater toxicity (side effects).

DETAILED DESCRIPTION:
Brain metastases are the most common intracranial tumors and occur in approximately 25% of patients with cancer. In the US, approximately 170,000 cancer patients a year are diagnosed with brain metastases.

The prognosis of patients with brain metastases is variable and depends on several factors, including performance status, age, control of the primary tumor, and extent of extracranial disease. Historically, patients with brain metastases who receive supportive care only have median survival of 1 to 2 months. However, a subgroup of patients with favorable prognosis who undergo treatment can enjoy an extended life expectancy with median survival of 10 to 16 months. Treatment options for brain metastases include medical management, surgery, and radiation therapy (radiotherapy). Both surgery and radiotherapy have an important role in management of brain metastases, and an optimized treatment plan may include both. It is well-established that surgery followed by conventional whole brain radiation (WBRT) decreases local recurrence and improves median survival compared to WBRT alone. Conventional WBRT is administered as radiotherapy to the whole cranium delivered in 10 to 20 daily treatments.

For this study, radiotherapy will be delivered using stereotactic radiosurgery (SRS) to treat individual metastases. SRS has the advantage of sparing normal brain tissue. In SRS, high energy radiation is precisely directed at the target lesion. Due to the steep fall-off of the radiation dose away from the target, the advantage of relative sparing of the normal brain may be realized. The present study is based on a rationale of treating brain metastases with surgical resection followed by adjuvant SRS to the resection cavity, while deferring conventional WBRT for salvage therapy.

WBRT is associated with a short-term decline in quality of life and long-term deficits in neurocognitive function ("late effects"). Late toxicity of WBRT, such as memory impairment and dementia, is usually irreversible and is likely due to demyelination, vascular damage, and necrosis. Following WBRT, the actuarial rate of neurocognitive toxicity at 2 years can be up to 49%. Recipients of WBRT may demonstrate a > 2 standard deviation decline in their performance at 6 months. Compared to SRS alone, WBRT was reported to be associated with a marked decline in learning and memory function at 4 months (49% vs 23%, in favor of SRS).

To minimize the potential late effects of WBRT, investigators have explored the use of SRS alone, deferring the use of WBRT for salvage treatment if needed. Both retrospective analyses and a prospective randomized trial reported no apparent survival benefit to combining WBRT with SRS compared to SRS alone

Primary Objectives: Determine the maximum tolerated dose (MTD) of stereotactic radiosurgery (SRS).

Secondary Objectives:

1. Determine the local control rate as assessed on MRI and clinical exam.
2. Determine short- and long-term adverse effects.
3. Determine the distant intra-cranial control rate.
4. Determine the overall survival rate.
5. Assess the patient's health related quality of life.

Treatment Group assignment will be by SRS dose level. SRS will be administered as 3 fractions. Radiation dose is administered as "Greys" (or "Grays"; abbreviated Gy), a unit by which radiation is measured. Treatment Groups are as follows: Group 1 = 24 Gy (administered as 8 Gy x 3) Group 2 = 7 Gy (9 Gy x 3); Group 3 = 30 Gy (10 Gy x 3); Group 4 = 33 Gy (11 Gy x 3).

Within each Treatment Group, analysis may be stratified by tumor size and suitability for surgical resection, as below. For those participants eligible for surgical resection, the procedure will be conducted in advance of the SRS treatment.

* Strata A will be those with tumors 4.2 to 14.1 cm³, and suitable for resection.
* Strata B will be those with tumors 4.2 to 14.1 cm³, but not suitable for resection.
* Strata C will be those with tumors 14.2 to 33.5 cm³, and suitable for resection.
* Strata D will be those with tumors 14.2 to 33.5 cm³, but not suitable for resection.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 18 years and older
* Pathologically-proven solid tumor malignancy
* 1 to 4 brain metastases, one of which is 4.2 to 33.5 cm³.
* Prior surgery or SRS is allowed as long as the target metastatic lesion in this study has not previously been treated with SRS.
* Prior cytotoxic systemic therapy must be completed ≥ 5 days prior to radiosurgery. No concurrent cytotoxic systemic therapy along with SRS. Cytotoxic systemic therapy to start ≥ 5 days after the completion of SRS.
* Life expectancy of ≥ 12 weeks.
* Ability to understand and the willingness to sign a written informed consent.

EXCLUSION CRITERIA

* Previously treated with whole brain irradiation
* Target metastatic lesion previously been treated with SRS.
* > 4 total brain metastases at the time of initial evaluation.
* Pregnant
* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Choi, Principal Investigator — Stanford University; Scott Soltys, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahimy E, Dudley SA, von Eyben R, Pollom EL, Seiger K, Modlin L, Wynne J, Fujimoto D, Jacobs LR, Chang SD, Gibbs IC, Hancock SL, Adler JR, Li G, Choi CYH, Soltys SG. Phase I/II Dose-Escalation Trial of 3-Fraction Stereotactic Radiosurgery for Resection Cavities From Large Brain Metastases: Health-related Quality of Life Outcomes. Am J Clin Oncol. 2021 Nov 1;44(11):588-595. doi: 10.1097/COC.0000000000000868. PMID 34670228

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Started | 20 | 12 | 12 | 12
Strata A: Small Tumor, Resected | 6 | 6 | 6 | 6
Strata B: Small Tumor, Not Resected | 5 | 0 | 0 | 0
Strata C: Large Tumor, Resected | 8 | 6 | 6 | 6
Strata D: Large Tumor, Not Resected | 1 | 0 | 0 | 0
Completed | 20 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS | Total
Number analyzed (Participants) | 20 | 12 | 12 | 12 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 5 | 7 | 7 | 35
  >=65 years | 4 | 7 | 5 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.0) | 67.2 (12.0) | 58.9 (12.2) | 59.2 (12.1) | 61.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 6 | 24
  Male | 12 | 7 | 7 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 2 | 6
  Not Hispanic or Latino | 15 | 6 | 10 | 10 | 41
  Unknown or Not Reported | 4 | 5 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 5 | 11 | 11 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 0 | 1 | 14
Region of Enrollment [Number; unit: participants]
  United States | 20 | 12 | 12 | 12 | 56

OUTCOME MEASURES:

1. Primary Outcome: Stereotactic Radiosurgery (SRS) Maximum-tolerated Dose (MTD)
Description: The maximum-tolerated Dose (MTD) of stereotactic radiosurgery (SRS) was assessed based on the number of dose-limiting toxicities (DLTs). DLT was defined as any treatment-related grade 3, 4, or 5 central nervous system (CNS) radiation morbidity observed within 30 days of radiosurgery. CNS radiation morbidity was further defined as.
  * 5 = Death
  * 4 = Serious neurologic impairment such as paralysis, coma, or seizures > 3/week
  * 3 = Neurologic findings requiring hospitalization
  * 2 = Neurologic findings present sufficient to require attendant care
  * 1 = Fully functional status (ie, able to work) with minor neurologic findings; no medication needed
  * 0 = No Change
  The outcome is expressed as number of DLTs experienced by participants, by radiotherapy dose cohort and tumor size, a number without dispersion. Per protocol, the MTD of SRS was defined as either the dose level below that at which 4+ DLTs were experienced by 12 subjects, or the maximum dose administered without MTD.
Time Frame: 60 days
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS).
Measure: Number; unit: Dose-limited toxicity (DLT) events
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 20 | 12 | 12 | 12
Dose-limited toxicity (DLT) events
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 6 | 6
  Strata A: Small tumor, resected | 0 | 0 | 0 | 0
  Strata B: Small tumor, not resected: number analyzed (Participants) | 5 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 0 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 8 | 6 | 6 | 6
  Strata C: Large tumor, resected | 0 | 0 | 0 | 0
  Strata D: Large tumor, not resected: number analyzed (Participants) | 1 | 0 | 0 | 0
  Strata D: Large tumor, not resected | 0 |  |  |

2. Secondary Outcome: Local Disease Control
Description: Local disease control (treatment response) was assessed on the basis of tumor size before and 12 months after treatment. Treatment response was based on the following criteria. Tumor area is determined as the product of 2 measurements of lesion diameter.
  * Complete response (CR): The tumor is no longer seen within the radiosurgical target volume
  * Partial response (PR): Decrease of > 50% in tumor area
  * Minor response (MR): Decrease of < 50% in tumor area
  * Stable disease (SD): The scan shows no change.
  * Progression (P): A > 25% increase in tumor area, or any new lesion within the radiosurgical target volume.
  Local control is defined as as any treatment response other than progression. The outcome is as the number of participants that did not progress, by radiotherapy dose cohort and tumor size, a number without dispersion.
Time Frame: 12 months
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS). Only participants with 12-month treatment response data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 11 | 10 | 12 | 12
Participants
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 5 | 6
  Strata A: Small tumor, resected | 4 | 6 | 5 | 6
  Strata B: Small tumor, not resected: number analyzed (Participants) | 2 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 0 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 5 | 4 | 6 | 6
  Strata C: Large tumor, resected | 5 | 4 | 6 | 4
  Strata D: Large tumor, not resected: number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Distant Intra-cranial Disease Control
Description: Distant treatment failure (failure to achieve or maintain disease control) is defined as the radiographic appearance of a new or enhancing lesion more than 5 mm from the radiosurgical target volume. The outcome is expressed as the number of participants who have distant treatment failure after radiotherapy dose cohort and tumor size, a number without dispersion.
Time Frame: 12 months
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS). Only participants with 12-month disease status data are included.
Measure: Number; unit: participants
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 11 | 10 | 9 | 12
participants
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 5 | 6
  Strata A: Small tumor, resected | 4 | 3 | 2 | 2
  Strata B: Small tumor, not resected: number analyzed (Participants) | 2 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 2 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 5 | 4 | 4 | 6
  Strata C: Large tumor, resected | 3 | 3 | 3 | 3
  Strata D: Large tumor, not resected: number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Adverse Effects Within 30 Days
Description: Short-term adverse effects are defined as any adverse event related to the stereotactic radiosurgery (SRS), and occurring within 30 days of SRS. The outcome is expressed as the number of events experienced by participants, by radiotherapy dose cohort and tumor size, a number without dispersion.
Time Frame: 30 days
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS).
Measure: Number; unit: adverse events
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 20 | 12 | 12 | 12
adverse events
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 6 | 6
  Strata A: Small tumor, resected | 3 | 4 | 4 | 2
  Strata B: Small tumor, not resected: number analyzed (Participants) | 5 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 3 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 8 | 6 | 6 | 6
  Strata C: Large tumor, resected | 4 | 2 | 2 | 3
  Strata D: Large tumor, not resected: number analyzed (Participants) | 1 | 0 | 0 | 0
  Strata D: Large tumor, not resected | 1 |  |  |

5. Secondary Outcome: Adverse Effects More Than 30 Days up to 1 Year
Description: Long-term adverse effects are defined as any adverse event related to the stereotactic radiosurgery (SRS), and occurring more 30 days but within 12 months of SRS. The outcome is expressed as the number of events experienced by participants, by radiotherapy dose cohort and tumor size, a number without dispersion.
Time Frame: after 30 days and up to 1 year
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS). Only participants surviving more than 30 days are included.
Measure: Number; unit: adverse events
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 19 | 12 | 12 | 12
adverse events
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 6 | 6
  Strata A: Small tumor, resected | 6 | 1 | 3 | 2
  Strata B: Small tumor, not resected: number analyzed (Participants) | 5 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 1 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 8 | 6 | 6 | 6
  Strata C: Large tumor, resected | 3 | 4 | 6 | 5
  Strata D: Large tumor, not resected: number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is assessed as remaining alive 3 years after stereotactic radiosurgery (SRS) therapy. The outcome is expressed as the number of participants alive 3 years after SRS, by radiotherapy dose cohort and tumor size, a number without dispersion.
Time Frame: 3 years
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 20 | 12 | 12 | 12
Participants
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 6 | 6
  Strata A: Small tumor, resected | 3 | 4 | 3 | 5
  Strata B: Small tumor, not resected: number analyzed (Participants) | 5 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 2 |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 8 | 6 | 6 | 6
  Strata C: Large tumor, resected | 5 | 2 | 4 | 2
  Strata D: Large tumor, not resected: number analyzed (Participants) | 1 | 0 | 0 | 0
  Strata D: Large tumor, not resected | 0 |  |  |

7. Secondary Outcome: Health-related Quality of Life (HR-QoL), as Measured by EORTC QLQ-C30
Description: Health-related quality of life (HR-QoL), was assessed based on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients (QLQ-C30) survey, a survey of 28 questions with the following responses / numerical values.
  1. Not at all
  2. A Little
  3. Quite a Bit
  4. Very Much Response range is 28 to 112, normalized to a 100 point scale. Lower values indicate little effect of disease, and higher values indicate greater effect. The outcome is expressed as the median value with full range, by radiotherapy dose cohort and tumor size.
Time Frame: 6 months
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS). Only participants providing 6-month European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients (QLQ-C30) health-related quality of life (HR-QoL) data are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 15 | 11 | 6 | 12
score on a scale
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 5 | 6
  Strata A: Small tumor, resected | 100 [58.3 to 100] | 83.3 [16.7 to 100] | 75 [16.7 to 100] | 50 [33.3 to 100]
  Strata B: Small tumor, not resected: number analyzed (Participants) | 3 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 75 [66.7 to 87.3] |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 6 | 5 | 1 | 6
  Strata C: Large tumor, resected | 87.5 [83.3 to 96.7] | 75 [25 to 100] | 83.3 [83.3 to 83.3] | 83.3 [58.33 to 83.3]
  Strata D: Large tumor, not resected: number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Health-related Quality of Life (HR-QoL), as Measured by EORTC Brain Cancer Module QLQ-BN20
Description: Health-related quality of life (HR-QoL), was assessed based on the European Organisation for Research and Treatment of Cancer (EORTC) Brain Cancer Module (QLQ-BN20), a survey of 20 questions with the following responses / numerical values.
  1. Not at all
  2. A Little
  3. Quite a Bit
  4. Very Much Response range is 20 to 80, normalized to a 0 to 100 scale. Lower values indicate little effect of disease, and higher values indicate greater effect. The outcome is expressed as the median value with full range, by radiotherapy dose cohort and tumor size.
Time Frame: 6 months
Population: There were few participants who did not receive tumor resection, and these were restricted to Arm 1 (24 Grey SRS). Only participants with 6-month European Organisation for Research and Treatment of Cancer (EORTC) Brain Cancer Module (QLQ-BN20) health-related quality of life (HR-QoL) data are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
Number analyzed (Participants) | 16 | 11 | 6 | 12
score on a scale
  Strata A: Small tumor, resected: number analyzed (Participants) | 6 | 6 | 5 | 6
  Strata A: Small tumor, resected | 0 [0 to 8.3] | 16.7 [0 to 75] | 16.5 [0 to 33.3] | 16.7 [0 to 25]
  Strata B: Small tumor, not resected: number analyzed (Participants) | 2 | 0 | 0 | 0
  Strata B: Small tumor, not resected | 0 [0 to 0] |  |  |
  Strata C: Large tumor, resected: number analyzed (Participants) | 8 | 5 | 1 | 6
  Strata C: Large tumor, resected | 12.5 [8.3 to 33.3] | 33.3 [0 to 83.3] | 8.3 [0 to 16.7] | 8.3 [0 to 16.7]
  Strata D: Large tumor, not resected: number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm 1 - 24 Grey SRS | Arm 2 - 27 Grey SRS | Arm 3 - 30 Grey SRS | Arm 4 - 33 Grey SRS
All-Cause Mortality (participants affected / at risk) | 10/20 | 6/12 | 5/12 | 5/12
Serious Adverse Events (participants affected / at risk) | 13/20 | 6/12 | 12/12 | 3/12
Other Adverse Events (participants affected / at risk) | 20/20 | 12/12 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - 24 Grey SRS (N=20) | Arm 2 - 27 Grey SRS (N=12) | Arm 3 - 30 Grey SRS (N=12) | Arm 4 - 33 Grey SRS (N=12)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal and urinary disorders -Others, Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders-Others, retrosigmoid stent migration to colon wall (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Altered mental status (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain-leg pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified-Other disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Death NOS (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Infection and infectations-other, fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - 24 Grey SRS (N=20) | Arm 2 - 27 Grey SRS (N=12) | Arm 3 - 30 Grey SRS (N=12) | Arm 4 - 33 Grey SRS (N=12)
Allopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ear and labyrinth disorders-Other, imbalance (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 5 (5)
Eye disorders - Other, diplopia (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eye disorders - Other, visual field loss (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT00928226/Prot_SAP_000.pdf